CLINICAL TRIAL: NCT01211197
Title: Relative Bioavailability of a 12.5 mg BI 10773 / 1000 mg Metformin Fixed Dose Combination Tablet Compared With Its Monocomponents and Administered With and Without Food (an Open-label, Randomised, Single-dose, Three-way Crossover, Phase I Trial in Healthy Volunteers)
Brief Title: Bioavailability of a Fixed Dose Combination Tablet With Empagliflozin (BI 10773) and Metformin Compared With the Monocomponents and Effect of Food on Bioavailability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1276.5; 2010-018589-22 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Results first posted 2015-08-21 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

ARMS (3):
- A (Experimental): 3 treatments will be investigated in randomized order
  Interventions: Drug: A: BI 10773 / metformin tablet
- B (Experimental): 3 treatments will be investigated in randomized order
  Interventions: Drug: B: BI 10773 tablet and metformin tablet
- C (Experimental): 3 treatments will be investigated in randomized order
  Interventions: Drug: C: BI 10773 / metformin tablet

INTERVENTIONS:
Drug: C: BI 10773 / metformin tablet — BI 10773 / metformin fixed dose combination tablet after a high fat, high caloric meal
  Arms: C
Drug: B: BI 10773 tablet and metformin tablet — BI 10773 and metformin single tablets, administered together in fasted state
  Arms: B
Drug: A: BI 10773 / metformin tablet — BI 10773 / metformin fixed dose combination tablet in fasted state
  Arms: A

SUMMARY:
The objective of the current study is to determine the relative bioavailability of a BI 10773 / metformin fixed dose combination tablet compared to single tablets of BI 10773 and metformin when administered together and to assess the effect of food on the bioavailability the fixed dose combination tablet

ELIGIBILITY:
Inclusion criteria:

1. Healthy males and females according to the following criteria
2. Body Mass Index 18.5 to 29.9 kg/m2 (incl.)

Exclusion criteria:

1. Any finding of the medical examination (including Blood Pressure, Pulse Rate and electrocardiogram) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1276.5.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An open label, randomised, three-way crossover study. A washout period of at least 7 days was respected between drug administrations.
Groups:
- FDC Fasted / Individual Tablets Fasted / FDC Fed: Patients received the three treatments in the following order:
  * FDC tablet, containing 12.5mg empagliflozin (BI 10773) and 1000mg metformin, under fasted conditions
  * 12.5mg empa and 1000mg metformin individual-component tablets under fasted conditions
  * FDC tablet, containing 12.5mg empagliflozin and 1000mg metformin, under fed conditions
- FDC Fasted / FDC Fed / Individual Tablets Fasted: Patients received the three treatments in the following order:
  * FDC tablet, containing 12.5mg empagliflozin and 1000mg metformin, under fasted conditions
  * FDC tablet, containing 12.5mg empagliflozin and 1000mg metformin, under fed conditions
  * 12.5mg empa and 1000mg metformin individual-component tablets under fasted conditions
- Individual Tablets Fasted / FDC Fasted / FDC Fed: Patients received the three treatments in the following order:
  * 12.5mg empa and 1000mg metformin individual-component tablets under fasted conditions
  * FDC tablet, containing 12.5mg empagliflozin and 1000mg metformin, under fasted conditions
  * FDC tablet, containing 12.5mg empagliflozin and 1000mg metformin, under fed conditions
- Individual Tablets Fasted / FDC Fed / FDC Fasted: Patients received the three treatments in the following order:
  * 12.5mg empa and 1000mg metformin individual-component tablets under fasted conditions
  * FDC tablet, containing 12.5mg empagliflozin and 1000mg metformin, under fed conditions
  * FDC tablet, containing 12.5mg empagliflozin and 1000mg metformin, under fasted conditions
- FDC Fed / FDC Fasted / Individual Tablets Fasted: Patients received the three treatments in the following order:
  * FDC tablet, containing 12.5mg empagliflozin and 1000mg metformin, under fed conditions
  * FDC tablet, containing 12.5mg empagliflozin and 1000mg metformin, under fasted conditions
  * 12.5mg empa and 1000mg metformin individual-component tablets under fasted conditions
- FDC Fed / Individual Tablets Fasted / FDC Fasted: Patients received the three treatments in the following order:
  * FDC tablet, containing 12.5mg empagliflozin and 1000mg metformin, under fed conditions
  * 12.5mg empa and 1000mg metformin individual-component tablets under fasted conditions
  * FDC tablet, containing 12.5mg empagliflozin and 1000mg metformin, under fasted conditions
Period: Treatment Period 1 (1 Day)
Arm/Group | FDC Fasted / Individual Tablets Fasted / FDC Fed | FDC Fasted / FDC Fed / Individual Tablets Fasted | Individual Tablets Fasted / FDC Fasted / FDC Fed | Individual Tablets Fasted / FDC Fed / FDC Fasted | FDC Fed / FDC Fasted / Individual Tablets Fasted | FDC Fed / Individual Tablets Fasted / FDC Fasted
Started | 3 | 3 | 3 | 3 | 2 | 2
Completed | 3 | 3 | 3 | 3 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1 (7 Days)
Arm/Group | FDC Fasted / Individual Tablets Fasted / FDC Fed | FDC Fasted / FDC Fed / Individual Tablets Fasted | Individual Tablets Fasted / FDC Fasted / FDC Fed | Individual Tablets Fasted / FDC Fed / FDC Fasted | FDC Fed / FDC Fasted / Individual Tablets Fasted | FDC Fed / Individual Tablets Fasted / FDC Fasted
Started | 3 | 3 | 3 | 3 | 2 | 2
Completed | 3 | 3 | 2 | 3 | 2 | 2
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Period: Treatment Period 2 (1 Day)
Arm/Group | FDC Fasted / Individual Tablets Fasted / FDC Fed | FDC Fasted / FDC Fed / Individual Tablets Fasted | Individual Tablets Fasted / FDC Fasted / FDC Fed | Individual Tablets Fasted / FDC Fed / FDC Fasted | FDC Fed / FDC Fasted / Individual Tablets Fasted | FDC Fed / Individual Tablets Fasted / FDC Fasted
Started | 3 | 3 | 2 | 3 | 2 | 2
Completed | 3 | 3 | 2 | 3 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (7 Days)
Arm/Group | FDC Fasted / Individual Tablets Fasted / FDC Fed | FDC Fasted / FDC Fed / Individual Tablets Fasted | Individual Tablets Fasted / FDC Fasted / FDC Fed | Individual Tablets Fasted / FDC Fed / FDC Fasted | FDC Fed / FDC Fasted / Individual Tablets Fasted | FDC Fed / Individual Tablets Fasted / FDC Fasted
Started | 3 | 3 | 2 | 3 | 2 | 2
Completed | 2 | 3 | 2 | 3 | 2 | 2
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (1 Day)
Arm/Group | FDC Fasted / Individual Tablets Fasted / FDC Fed | FDC Fasted / FDC Fed / Individual Tablets Fasted | Individual Tablets Fasted / FDC Fasted / FDC Fed | Individual Tablets Fasted / FDC Fed / FDC Fasted | FDC Fed / FDC Fasted / Individual Tablets Fasted | FDC Fed / Individual Tablets Fasted / FDC Fasted
Started | 2 | 3 | 2 | 3 | 2 | 2
Completed | 2 | 3 | 2 | 3 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Overall: An open label, randomised, three-way crossover study. The three treatments administered were
  * Fixed dose combination (FDC) tablet, containing 12.5mg empagliflozin and 1000mg metformin, under fasted conditions
  * 12.5mg empa and 1000mg metformin individual-component tablets under fasted conditions
  * Fixed dose combination (FDC) tablet, containing 12.5mg empagliflozin and 1000mg metformin, under fed conditions
  A washout period of at least 7 days was respected between drug administrations.
Arm/Group | Study Overall
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Empa: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of empagliflozin (empa) in plasma over the time interval from 0 extrapolated to infinity.
  Note the standard deviation is actually the coefficient of variation (CV).
Time Frame: 1 hour (h) before drug administration and 20 minutes (min), 40min, 1 h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 34h, 48h, 72h after drug administration
Population: Pharmacokinetic (PK) set included all evaluable subjects who took at least 1 dose of investigational medication, provided at least one observation for at least one primary PK endpoint without important protocol violations relevant to the evaluation of pharmacokinetics.
Measure: Mean (Standard Deviation); unit: nmol*h/L
Groups:
- FDC Fasted: A single fixed dose combination (FDC) tablet, containing 12.5mg empagliflozin and 1000mg metformin, under fasted conditions.
- Individual Tablets Fasted: 12.5mg empa and 1000mg metformin individual-component tablets under fasted conditions.
- FDC Fed: A single fixed dose combination (FDC) tablet, containing 12.5mg empagliflozin and 1000mg metformin, under fed conditions.
Arm/Group | FDC Fasted | Individual Tablets Fasted | FDC Fed
Number analyzed (Participants) | 15 | 16 | 14
nmol*h/L | 2920 (16.2) | 2860 (18.5) | 2710 (15.0)
Statistical Analysis 1: Comparison: FDC Fasted vs Individual Tablets Fasted; Ratio calculated as FDC fasted divided by individual tablets fasted; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric mean ratio = 100.59, 90% CI 2-sided [95.75 to 105.67], Standard Deviation 7.6 — Standard deviation is actually the intra-individual geometric coefficient of variation (gCV)
Statistical Analysis 2: Comparison: FDC Fasted vs FDC Fed; Ratio calculated as FDC fed divided by FDC fasted; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric mean ratio = 94.94, 90% CI 2-sided [89.85 to 100.33], Standard Deviation 8.0 — Standard deviation is actually the intra-individual gCV

2. Primary Outcome: Empa: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of empagliflozin (empa) in plasma.
  Note the standard deviation is actually the CV.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | FDC Fasted | Individual Tablets Fasted | FDC Fed
Number analyzed (Participants) | 15 | 16 | 14
nmol/L | 404 (17.4) | 405 (15.8) | 259 (20.3)
Statistical Analysis 1: Comparison: FDC Fasted vs Individual Tablets Fasted; Ratio calculated as FDC fasted divided by individual tablets fasted; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric mean ratio = 99.31, 90% CI 2-sided [91.76 to 107.49], Standard Deviation 12.2 — Standard deviation is actually the intra-individual gCV
Statistical Analysis 2: Comparison: FDC Fasted vs FDC Fed; Ratio calculated as FDC fed divided by FDC fasted; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric mean ratio = 64.30, 90% CI 2-sided [55.97 to 73.87], Standard Deviation 20.6 — Standard deviation is actually the intra-individual gCV

3. Secondary Outcome: Empa: Area Under the Curve 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of empagliflozin (empa) in plasma over the time interval from 0 to the time of the last quantifiable data point.
  Note the standard deviation is actually the CV.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol*h/L
Arm/Group | FDC Fasted | Individual Tablets Fasted | FDC Fed
Number analyzed (Participants) | 15 | 16 | 14
nmol*h/L | 2860 (16.3) | 2800 (18.6) | 2640 (15.1)
Statistical Analysis 1: Comparison: FDC Fasted vs Individual Tablets Fasted; Ratio calculated as FDC fasted divided by individual tablets fasted; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric mean ratio = 100.94, 90% CI 2-sided [96.03 to 106.11], Standard Deviation 7.7 — Standard deviation is actually the intra-individual gCV
Statistical Analysis 2: Comparison: FDC Fasted vs FDC Fed; Ratio calculated as FDC fed divided by FDC fasted; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric mean ratio = 94.39, 90% CI 2-sided [89.22 to 99.87], Standard Deviation 8.2 — Standard deviation is actually the intra-individual gCV

4. Secondary Outcome: Metformin: Area Under the Curve 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of metformin in plasma over the time interval from 0 to the time of the last quantifiable data point.
  Note the standard deviation is actually the CV.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | FDC Fasted | Individual Tablets Fasted | FDC Fed
Number analyzed (Participants) | 15 | 16 | 14
ng*h/mL | 9900 (17.9) | 9720 (22.3) | 9550 (19.7)
Statistical Analysis 1: Comparison: FDC Fasted vs Individual Tablets Fasted; Ratio calculated as FDC fasted divided by individual tablets fasted; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric mean ratio = 103.13, 90% CI 2-sided [95.59 to 111.25], Standard Deviation 11.7 — Standard deviation is actually the intra-individual gCV
Statistical Analysis 2: Comparison: FDC Fasted vs FDC Fed; Ratio calculated as FDC fed divided by FDC fasted; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric mean ratio = 96.96, 90% CI 2-sided [87.23 to 107.78], Standard Deviation 15.5 — Standard deviation is actually the intra-individual gCV

5. Primary Outcome: Metformin: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of metformin in plasma over the time interval from 0 extrapolated to infinity.
  Note the standard deviation is actually the CV.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | FDC Fasted | Individual Tablets Fasted | FDC Fed
Number analyzed (Participants) | 15 | 16 | 14
ng*h/mL | 10300 (16.9) | 10100 (21.2) | 10200 (15.6)
Statistical Analysis 1: Comparison: FDC Fasted vs Individual Tablets Fasted; Ratio calculated as FDC fasted divided by individual tablets fasted; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric mean ratio = 102.15, 90% CI 2-sided [93.87 to 111.15], Standard Deviation 13.0 — Standard deviation is actually the intra-individual gCV
Statistical Analysis 2: Comparison: FDC Fasted vs FDC Fed; Ratio calculated as FDC fed divided by FDC fasted; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric mean ratio = 100.67, 90% CI 2-sided [91.70 to 110.51], Standard Deviation 13.7 — Standard deviation is actually the intra-individual gCV

6. Primary Outcome: Metformin: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of metformin in plasma.
  Note the standard deviation is actually the CV.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | FDC Fasted | Individual Tablets Fasted | FDC Fed
Number analyzed (Participants) | 15 | 16 | 14
ng/mL | 1550 (19.1) | 1530 (23.4) | 1180 (25.5)
Statistical Analysis 1: Comparison: FDC Fasted vs Individual Tablets Fasted; Ratio calculated as FDC fasted divided by individual tablets fasted; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric mean ratio = 103.49, 90% CI 2-sided [95.30 to 112.39], Standard Deviation 12.7 — Standard deviation is actually the intra-individual gCV
Statistical Analysis 2: Comparison: FDC Fasted vs FDC Fed; Ratio calculated as FDC fed divided by FDC fasted; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric mean ratio = 75.13, 90% CI 2-sided [63.68 to 88.64], Standard Deviation 24.5 — Standard deviation is actually the intra-individual gCV

7. Secondary Outcome: Time to Maximum Measured Concentration (Tmax)
Description: Time from dosing to the maximum concentration of the analyte in plasma.
  Note the standard deviation is actually the CV.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | FDC Fasted | Individual Tablets Fasted | FDC Fed
Number analyzed (Participants) | 15 | 16 | 14
hours
  Tmax of empagliflozin | 1.50 (34.2) [0.67 to 2.50] | 1.75 (27.1) [1.00 to 2.50] | 3.00 (54.6) [1.00 to 8.00]
  Tmax of metformin | 2.50 (20.9) [2.00 to 4.00] | 2.50 (26.3) [1.50 to 4.00] | 3.00 (49.8) [1.50 to 8.00]

8. Secondary Outcome: Terminal Elimination Rate Constant in Plasma (λz)
Description: Terminal elimination rate constant in plasma.
  Note the standard deviation is actually the CV.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | FDC Fasted | Individual Tablets Fasted | FDC Fed
Number analyzed (Participants) | 15 | 16 | 14
1/h
  λz of empagliflozin | 0.0559 (43.9) | 0.0601 (53.2) | 0.0498 (46.6)
  λz of metformin | 0.0822 (73.3) | 0.0756 (82.7) | 0.0590 (108)

9. Secondary Outcome: Terminal Half-life in Plasma (T1/2)
Description: Terminal half-life of the analyte in plasma.
  Note the standard deviation is actually the CV.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | FDC Fasted | Individual Tablets Fasted | FDC Fed
Number analyzed (Participants) | 15 | 16 | 14
hours
  T1/2 of empagliflozin | 15.1 (46.6) | 16.0 (61.3) | 16.7 (43.0)
  T1/2 of metformin | 16.6 (94.6) | 17.8 (76.9) | 30.5 (89.0)

10. Secondary Outcome: Mean Residence Time in the Body After Oral Administration (MRTpo)
Description: Mean residence time of the analyte in the body after oral administration.
  Note the standard deviation is actually the CV.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | FDC Fasted | Individual Tablets Fasted | FDC Fed
Number analyzed (Participants) | 15 | 16 | 14
hours
  MRTpo of empagliflozin | 10.5 (17.6) | 10.9 (25.1) | 13.9 (23.0)
  MRTpo of metformin | 9.53 (52.0) | 10.2 (52.1) | 19.4 (101)

11. Secondary Outcome: Apparent Clearance After Extravascular Administration (CL/F)
Description: Apparent clearance of the analyte in the plasma after extravascular administration.
  Note the standard deviation is actually the CV.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | FDC Fasted | Individual Tablets Fasted | FDC Fed
Number analyzed (Participants) | 15 | 16 | 14
mL/min
  CL/F of empagliflozin | 162 (15.0) | 166 (17.1) | 174 (13.3)
  CL/F of metformin | 1670 (20.2) | 1730 (25.4) | 1670 (18.8)

12. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase (Vz/F)
Description: Apparent volume of distribution during the terminal phase (λz).
  Note the standard deviation is actually the CV.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | FDC Fasted | Individual Tablets Fasted | FDC Fed
Number analyzed (Participants) | 15 | 16 | 14
Litres
  Vz/F of empagliflozin | 210 (45.3) | 222 (58.0) | 250 (44.3)
  Vz/F of metformin | 2410 (99.5) | 2650 (86.0) | 4670 (112)

13. Secondary Outcome: Clinically Relevant Abnormalities for Physical Examination, Vital Signs, ECG, Blood Chemistry and Assessment of Tolerability by the Investigator.
Description: Clinically relevant abnormalities for physical examination, vital signs, ECG, blood chemistry and assessment of tolerability by the investigator. New abnormal findings or worsening of baseline conditions were reported as adverse events.
Time Frame: Drug administration up to 7 days after last drug administration, up to 8 days
Population: Treated set (TS) includes all subjects who took at least 1 dose of investigational medication and was used for safety analysis.
Measure: Number; unit: participants
Arm/Group | FDC Fasted | Individual Tablets Fasted | FDC Fed
Number analyzed (Participants) | 15 | 16 | 14
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Drug administration up to 7 days after last drug administration, up to 8 days
Groups:
- FDC Fed: A single fixed dose combination (FDC) tablet, containing 12.5mg empagliflozin and 1000mg metformin, under fasted conditions.
Arm/Group | FDC Fasted | Individual Tablets Fasted | FDC Fed
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 2/15 | 6/16 | 8/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FDC Fasted (N=15) | Individual Tablets Fasted (N=16) | FDC Fed (N=14)
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 3
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes